CLINICAL TRIAL: NCT05115435
Title: The Effect of Neuro Linguistic Programming on COVID-19 Fear in Kidney Transplant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Runida Dogan, Assistant Professor, Inonu University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: RDNLP
Record Dates: First submitted 2021-11-08; First posted 2021-11-10 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-11

CONDITIONS: Kidney Transplant Patients
Keywords: Neuro Linguistic Programming; fear of covid-19; kidney transplant patients; nurse
MeSH Terms: interventions — Neurolinguistic Programming

STUDY DESIGN:
Intervention Model Description: The population of the study consisted of patients who had kidney transplants in the hospital in question. The sample of the study was determined by power analysis. According to the calculation made using G*power 3.1 software, the sample size was determined as 74 (each group 37) with an effect size of 0.80, a margin of error of 0co.05, a confidence level of 0.95, and a population representation of 0.95. Simple random sampling method, one of the probability sampling methods, was used to determine the participants. Single-group columns between 1 and 300 were created using the Random Integer Generator method, which located in the Numbers sub-heading of the random.org website for the participants who met the sample selection criteria. Participants were randomly assigned to numbers 1 and 2, considering the numbers 1 and 2 in the column. The number of the experimental or control group was determined by drawing lots at the beginning of the research.
Who Masked: Participant
Masking Description: Participants did not know they were in the experimental or control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): No intervention was applied on the control group patients
- experimental group (Experimental): Sub modality Technique: People experience the world with their five senses, and the thoughts that an individual creates in his brain about a situation are coded with these five senses. When these encodings change, the individual's perception of the situation will also change
  Interventions: Behavioral: neuro linguistic programming

INTERVENTIONS:
Behavioral: neuro linguistic programming — Sub modality Technique: People experience the world with their five senses, and the thoughts that an individual creates in his brain about a situation are coded with these five senses. When these encodings change, the individual's perception of the situation will also change
  Arms: experimental group

SUMMARY:
The study was conducted experimentally to evaluate the effect of neurolinguistic programming on COVID-19 fear in kidney transplant patients.

DETAILED DESCRIPTION:
The study was conducted experimentally (prospective randomized single-blind clinical trial model) to evaluate the effect of neurolinguistic programming (NLP) on fear of Covid-19 in kidney transplant patients.

The study was carried out between June 2021 and October 2021. Personal Information Form and Fear of COVID-19 Scale (FCV-19S) were used to collect data. The data obtained from the research were evaluated with SPSS 25.

According to the calculation made using G*power 3.1 software, the sample size was determined as 74 (each group 37) with an effect size of 0.80, a margin of error of 0co.05, a confidence level of 0.95, and a population representation of 0.95. Simple random sampling method, one of the probability sampling methods, was used to determine the participants. Single-group columns between 1 and 300 were created using the Random Integer Generator method, which located in the Numbers sub-heading of the random.org website for the participants who met the sample selection criteria. Participants were randomly assigned to numbers 1 and 2, considering the numbers 1 and 2 in the column. The number of the experimental or control group was determined by drawing lots at the beginning of the research

ELIGIBILITY:
Inclusion Criteria:Patients who could communicate verbally, had no hearing problems, had a high or moderate fear of Covid-19 (20 or more), and had not applied NLP before were included in the study.

-

Exclusion Criteria: Patients who wanted to leave voluntarily at any stage after being included in the study, and who had to be hospitalized again for organ rejection or any other reason while the study was ongoing, were excluded from the study.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
A mean total score on the | Fear of COVID-19 Scale . After applying the personal information form and Fear of COVID-19 Scale (FCV-19S) to the patients in the experimental group, the sub-modality technique of NLP was applied once, and then FCV-19S was applied again one week later
  Fear of COVID-19 Scale (FCV-19S)

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - İnönü University, Malatya
  - İnönü Üniversitesi, Malatya

IPD SHARING:
Plan to Share IPD: Undecided
Data can be shared with the permission of the researchers.

REFERENCES:
- [Derived] Dogan A, Dogan R, Menekli T, Berktas HB. Effect of neuro-linguistic programming on COVID-19 fear in kidney transplant patients: A randomized controlled study. Complement Ther Clin Pract. 2022 Nov;49:101638. doi: 10.1016/j.ctcp.2022.101638. Epub 2022 Jul 4. PMID 35843115